CLINICAL TRIAL: NCT02389296
Title: The Forensic Psychiatric Nurse - Warden or Empathic Caregiver
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: HYMC-0021-15
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Psychiatric Nursing
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Forensic Psychiatric Nurses in Mental Health Centers: Psychiatric nurses working in forensic wards in mental health centers
  Interventions: Other: Questionnaire
- Psychiatric Nurses in General Hospitals: Psychiatric nurses working in general hospitals
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaires will be distributed to nursing staff

SUMMARY:
The aim of this study is to determine whether the work environment influences the role perception of nurses in psychiatric wards. This will be a comparative study. Questionnaires will be distributed to nurses working in psychiatric wards in 10 medical centers in Israel.

ELIGIBILITY:
Inclusion Criteria:

* RN Accredited Nurses
* Hebrew Speaking

Exclusion Criteria:

* Incomplete questionnaire

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Psychiatric nurses working in either general hospitals or in mental health centers in 10 medical centers in Israel.
Sampling Method: Probability Sample
Enrollment: 212 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Empathetic Caregiver | One year
  Questionnaire with Liekert Scale will determine nursing staff behavioral intention
Warden | One year
  Questionnaire with Liekert Scale will determine nursing staff behavioral intention